CLINICAL TRIAL: NCT06091527
Title: Treating Major Depression With Yoga Mono-therapy: 12-Week Randomized Controlled Trial
Brief Title: Treating Major Depression With Yoga Mono-therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-38755
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Depression Mild; Depression Moderate
Keywords: yoga; ayurveda; depression
MeSH Terms: conditions — Depression | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga practice (Experimental): Yoga practice groups
  Interventions: Behavioral: Yoga practice
- Education (Active Comparator): Education module group
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Yoga practice — 90-minute group yoga classes twice weekly for 12 weeks.
  Arms: Yoga practice
Behavioral: Education — 90-minute group education classes twice weekly for 12 weeks to learn holistic healthcare modules.
  Arms: Education

SUMMARY:
The goal of this single-center, single-blind, randomized, controlled, parallel group, interventional trial is to evaluate antidepressant efficacy of yoga monotherapy of 12-weeks duration in 180 adults meeting diagnostic criteria for mild-to-moderate major depression at the Zuckerberg San Francisco General Hospital. Researchers will compare the yoga interventions to an education control intervention on holistic healthcare.

DETAILED DESCRIPTION:
Consenting participants will be randomized equally to one of three in-person group interventions for 12 weeks: Standard yoga practice, Ayurvedic yoga practice, or educational attention-control modules. The primary outcome is depression severity, measured by Beck Depression Inventory-II (BDI) scores. Secondary outcomes include perceived stress, measured by Perceived Stress Scale (PSS) scores, and several biomarker assays associated with depression: methylation of the GrimAge epigenetic clock, nuclear factor kappa-B (NF-κB) transcription, leucocyte telomere length, interleukin-6 (IL-6) and brain-derived neurotropic factor (BDNF). Blinded assessors will conduct all outcome analyses at 12 weeks. The primary analysis will test whether the yoga groups combined achieve statistically greater change in BDI scores compared to the control group. Secondary analyses will test whether the yoga groups combined, compared to the control group, demonstrate statistically greater change in PSS scores and the aforementioned biomarker assays. In sub-analyses, investigators will assess whether Ayurvedic yoga participants, compared to Standard yoga participants, demonstrate statistically significant improvements in BDI scores, PSS scores, and depression biomarker assays over the 12-week intervention period.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Able to give voluntary, informed consent
* English-speaking
* Diagnosis of clinical depression

Exclusion criteria:

* Current use of antidepressant medication
* Current engagement in psychotherapy
* Current pregnancy
* Significant medical issues interfering with yoga practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory-II score | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks and 12 weeks
  The Beck Depression Inventory-II is one of the most commonly used instruments in psychiatric research; it has been translated and validated in many different languages, appearing in hundreds of studies worldwide. The Beck Depression Inventory-II is a 21-item validated instrument for the self-report of depressive symptoms; it can typically be completed in 5 minutes. Each item on the Beck Depression Inventory-II can be scored from 0 to 3, with the total score derived by summing the individual item scores. A total score of 14-19 suggests mild depression, 20-28 suggests moderate depression, and 29-63 suggests severe depression.

SECONDARY OUTCOMES:
Change in Perceived Stress Scale score | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks and 12 weeks
  The Perceived Stress Scale is a commonly used instrument in psychiatric research; it has been translated and in many different languages, appearing in hundreds of studies worldwide. The Perceived Stress Scale is a 10-item validated questionnaire used to assess stress levels in individuals. It can typically be completed in 5 minutes and evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month. Each item on the Perceived Stress Scale can be scored 0 to 4, with the total score derived by summing the individual item scores. Higher scores indicate higher levels of perceived stress and there are no score cut-offs published by the developer.
Change in methylation of the GrimAge epigenetic clock | Baseline and 12 weeks
  Blood samples will be drawn from each enrolled participant at the Baseline Visit and at 12 weeks.
Change in transcription of the nuclear factor kappa-B (NF-κB) pathway | Baseline and 12 weeks
  Blood samples will be drawn from each enrolled participant at the Baseline Visit and at 12 weeks.
Change in plasma interleukin-6 (IL-6) level | Baseline and 12 weeks
  Blood samples will be drawn from each enrolled participant at the Baseline Visit and at 12 weeks.
Change in telomere length of leukocytes | Baseline and 12 weeks
  Blood samples will be drawn from each enrolled participant at the Baseline Visit and at 12 weeks.
Change in plasma brain-derived neurotropic factor (BDNF) level | Baseline and 12 weeks
  Blood samples will be drawn from each enrolled participant at the Baseline Visit and at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Prathikanti, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prathikanti S, Rivera R, Cochran A, Tungol JG, Fayazmanesh N, Weinmann E. Treating major depression with yoga: A prospective, randomized, controlled pilot trial. PLoS One. 2017 Mar 16;12(3):e0173869. doi: 10.1371/journal.pone.0173869. eCollection 2017. PMID 28301561
- [Background] Wu Y, Yan D, Yang J. Effectiveness of yoga for major depressive disorder: A systematic review and meta-analysis. Front Psychiatry. 2023 Mar 23;14:1138205. doi: 10.3389/fpsyt.2023.1138205. eCollection 2023. PMID 37032928
- [Background] Naveen GH, Varambally S, Thirthalli J, Rao M, Christopher R, Gangadhar BN. Serum cortisol and BDNF in patients with major depression-effect of yoga. Int Rev Psychiatry. 2016 Jun;28(3):273-8. doi: 10.1080/09540261.2016.1175419. Epub 2016 May 13. PMID 27174729
- [Background] Deng W, Cheung ST, Tsao SW, Wang XM, Tiwari AF. Telomerase activity and its association with psychological stress, mental disorders, lifestyle factors and interventions: A systematic review. Psychoneuroendocrinology. 2016 Feb;64:150-63. doi: 10.1016/j.psyneuen.2015.11.017. Epub 2015 Nov 25. PMID 26677763
- [Background] Nugent NR, Brick L, Armey MF, Tyrka AR, Ridout KK, Uebelacker LA. Benefits of Yoga on IL-6: Findings from a Randomized Controlled Trial of Yoga for Depression. Behav Med. 2021 Jan-Mar;47(1):21-30. doi: 10.1080/08964289.2019.1604489. Epub 2019 May 29. PMID 31141465
- [Background] Pisanu C, Tsermpini EE, Skokou M, Kordou Z, Gourzis P, Assimakopoulos K, Congiu D, Meloni A, Balasopoulos D, Patrinos GP, Squassina A. Leukocyte telomere length is reduced in patients with major depressive disorder. Drug Dev Res. 2020 May;81(3):268-273. doi: 10.1002/ddr.21612. Epub 2019 Nov 1. PMID 31675136
- [Background] Protsenko E, Yang R, Nier B, Reus V, Hammamieh R, Rampersaud R, Wu GWY, Hough CM, Epel E, Prather AA, Jett M, Gautam A, Mellon SH, Wolkowitz OM. "GrimAge," an epigenetic predictor of mortality, is accelerated in major depressive disorder. Transl Psychiatry. 2021 Apr 6;11(1):193. doi: 10.1038/s41398-021-01302-0. PMID 33820909
- [Background] Tolahunase MR, Sagar R, Faiq M, Dada R. Yoga- and meditation-based lifestyle intervention increases neuroplasticity and reduces severity of major depressive disorder: A randomized controlled trial. Restor Neurol Neurosci. 2018;36(3):423-442. doi: 10.3233/RNN-170810. PMID 29614706
- [Background] Venditti S, Verdone L, Reale A, Vetriani V, Caserta M, Zampieri M. Molecules of Silence: Effects of Meditation on Gene Expression and Epigenetics. Front Psychol. 2020 Aug 11;11:1767. doi: 10.3389/fpsyg.2020.01767. eCollection 2020. PMID 32849047